CLINICAL TRIAL: NCT03313921
Title: The MORE Study: Manifest vs. Online Refraction Evaluation. A Clinical Validation of Online Refraction
Brief Title: The MORE Study: Manifest vs. Online Refraction Evaluation
Acronym: MORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Robert P.L. Wisse, MD PhD, Ophthalmologist, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL61478.041.17
Record Dates: First submitted 2017-09-21; First posted 2017-10-18 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Refraction Error; Myopia; Astigmatism
Keywords: myopia; astigmatism; online assessment; refractive error
MeSH Terms: conditions — Refractive Errors; Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: cross-sectional open-label non-inferiority assessment of a novel diagnostic entity compared to current gold-standard in two seperate groups of patients (healthy and diseased)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Manifest Refraction (Experimental): All participants will undergo three assessments of refractive error, in random order. All will perform an unsupervised manifest refraction with the use of a computer screen and their smartphone. Next, a regular manifest refraction assessment performed by an optometrist will function as active comparator. An automated refraction assessment will be performed to relate the quality and repeatability of the online refraction to another unsupervised method of refraction assessment.
  Interventions: Diagnostic Test: Online Manifest Refraction

INTERVENTIONS:
Diagnostic Test: Online Manifest Refraction — The online manifest refraction is performed with a web-based application and consists of an assessment of visual acuity, an assessment of spherical refractive error, and an assessment of cylinder refractive error. The software is a class 1 CE-approved medical device.
  The automated refraction is measured with a regular office-based autorefractor device; TOPCON RM-8000.
  Other Names: Easee online refraction

SUMMARY:
The assessment of the refractive state of the eye is a fundamental and important part of ophthalmic and optometric clinical practice. The development of an unsupervised online subjective refraction method makes a refraction more accessible and can be quite cost-saving.

In this study, the investigators want to validate an online refraction method which was recently created in the Netherlands. The study comprises two different set of participants: Part one contains fifty healthy volunteers, 18-40 years of age, with a refractive error and no other ophthalmic pathology. Part two contains fifty patients with an ophthalmic pathology.

The online refraction outcomes will be compared to a manifest refraction and automated refraction in a cross-sectional study design.

DETAILED DESCRIPTION:
Uncorrected refractive errors cause significant economic implications in both high and low income countries in terms of the loss of potential productivity (Williams et al. (2015)). The prevalence of uncorrected refractive errors is, despite of the available clinical services, still huge; visual impairment is in 42 percent of the cases the result of an uncorrected refractive error worldwide (Williams et al. (2015)). Even in high income countries, this issue remains prevalent. Therefore, the access to the available clinical services has to be simplified. The development of an online refraction method will make a refraction more accessible for patients and can be cost-saving. Clinicians can easily take an online method to places where it's needed for example in low income countries.

There are several methods to measure a refractive error. The 'golden standard' to prescribe spectacles is a manifest refraction (Thibos, Hong, Bradley & Applegate (2004)). This method was already described by F.C. Donders in 1864 and is performed with trial lenses and a visual acuity chart to measure the refraction error (Donders (1864)). An automated refraction is a quick routine machine based assessment, mainly used as a starting point for a manifest refraction and is based on retinoscopy (Nissman et al., (2004)).

At the moment, several online refraction methods are available. However, these methods are not scientifically validated, unavailable outside the United States of America (USA) or not designed for customers. One of these online refraction methods is Opternative (Opternative (2017)). Opternative is currently used in the USA and is still developing (Opternative (2017)). It's a self-directed online refraction method using a computer-based response to presented stimuli with the use of a smartphone and a computer. Another method is EyeNetra (EyeNetra (2017) & Ohlendorf, Leube & Wahl (2016)). The use of this method is limited due to the need of special equipment such as a portable autorefractor, an autolensometer and a phoropter. Therefore, EyeNetra is mainly designed for optometrists and ophthalmologists for low-income populations. The same applies to SVOne; this method uses a Hartmann-Shack wavefront aberrometer which the user can attach to a smartphone (Ohlendorf, Leube & Wahl (2016)). Other online refraction methods are 6over6, but this method has not been released yet (6over6, (2017)), and Warby Parker (Warby Parker, (2017)).

There are also online visual acuity tests to measure the visual acuity only. The mobile devices to test the visual acuity are PeekVision, 6over6, Opternative, Eyenetra and DigiSight (Ludwig et al., (2016)).

Currently, digitalization is affecting our way of life. Technology can be used to design products to easily determine if someone has a refractive error. This can, in the future, solve a big part of the problem of uncorrected refractive errors and the leading cause of blindness worldwide. The aim of this study is to validate a recently created online refraction method by comparing the outcomes of the online refraction method with the 'golden standard' manifest refraction.

ELIGIBILITY:
inclusion criteria:

1. Group one:

   * Age: 18-40 years
   * Master the Dutch language
   * Capable to perform the tests adequately.
2. Group two:

   * Age: 18-40 years
   * Master the Dutch language
   * Capable to perform the tests adequately.
   * Diagnosis of keratoconus.

Exclusion Criteria:

1. Group one:

   * No informed consent
   * Diabetes
   * Pregnancy or lactation
   * High hyperopia/myopia (>6D)
   * An ophthalmic history besides ametropia
2. Group two:

   * No informed consent
   * Diabetes
   * Pregnancy or lactation
   * High hyperopia/myopia (>6D)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Refractive error | All three measurements (automated refraction, manifest refraction and online refraction) will be performed subsequently on the same 1 day. Data collection will take place between november 2017 and january 2018. No follow up measurements are required.
  The refractive error is recorded in a Sphere power (D), a Cylinder power (D) and a Cylinder axis (°). These are converted into vectors by Fourier analysis.

SECONDARY OUTCOMES:
Maximum distance visual acuity | The visual acuity test will take place on the same 1 day as the other measurements. Data collection will take place between november 2017 and january 2018. No follow up measurements are required.
  The maximum visual acuity as assessed during the refraction procedure using an ETDRS visual acuity chart and converted into logMAR values.
Participant satisfaction | The questionnaire will be filled in on the same 1 day as the other measurements. Data collecting will take place between november 2017 and january 2018. No follow up measurements are required.
  Questionnaire on user experience of the smartphone application.
Telemetry | Measurements of the duration of the online test will happen 1 day during the online refraction test. Collecting data will take place between November 2017 and January 2018. No follow up measurements are required.
  Duration of the online test time

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wisse, MD PHD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wisse RPL, Muijzer MB, Cassano F, Godefrooij DA, Prevoo YFDM, Soeters N. Validation of an Independent Web-Based Tool for Measuring Visual Acuity and Refractive Error (the Manifest versus Online Refractive Evaluation Trial): Prospective Open-Label Noninferiority Clinical Trial. J Med Internet Res. 2019 Nov 8;21(11):e14808. doi: 10.2196/14808. PMID 31702560
- See also: website of the online refractive assessment — https://easee.online/